CLINICAL TRIAL: NCT03362073
Title: A Phase II Study About Efficacy and Safety of the Continuous IntraVenous Infusion of Ketamine in Terminally Ill Cancer Patients With Refractory Cancer Pain
Brief Title: Continuous IntraVenous Infusion of Ketamine in Terminally Ill Cancer Patients
Acronym: CIVIK
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kwonoh Park, MD phD, Professor, clinical research, Pusan National University Yangsan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIVIK
Record Dates: First submitted 2017-11-15; First posted 2017-12-05 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Ketamine; Refractory Cancer Pain
Keywords: Ketamine; Refractory cancer pain; Terminally ill cancer patients; Palliative care
MeSH Terms: conditions — Cancer Pain | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Prospective, Single institution, Open-label, Phase 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketamine (Experimental): continuous intravenous infusion of ketamine
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Application of ketamine using continuous intravenous infusion method during 5 days
  * Ketamine 100mg/2ml + 5% Dextrose water or Normal saline 98 ml mixed fluid
  * Dose schedule: 0.05mg/kg/hr -> 0.10mg/kg/hr -> … -> 0.5mg/kg/hr (increase dose at a rate of 0.05mg/kg/hr every 8 hours)

SUMMARY:
To establish the role of ketamine in hospitalized terminally ill cancer patients with refractory cancer pain, using continuous intravenous infusion of ketamine

DETAILED DESCRIPTION:
* There are approximately 20 percent patients of refractory cancer pain, which is troubled with uncontrolled pain though treatment including opioids.
* Ketamine has been showed the performance of Ketamine, N-methyl-D-aspartate (NMDA) receptor blocker, in refractory cancer pain based on prior studies.
* We cannot yet confirm the role of Ketamine comparing the benefit and risk due to incompatible results of prior studies. Additionally, most of prior studies were studied in heterogenous groups, which are from beginning of palliative chemotherapy to terminal status, so role of ketamine was not assessed in homogeneous terminally ill cancer patients. And they has used mostly 'bolus intravenous infusion' or 'continuous subcutaneous infusion (CSCI)', relatively rare in continuous intravenous infusion (CIVI).
* The bolus intravenous method is convenient but is concerned with leading to relatively severe adverse events due to poor general condition of terminally ill cancer patients, the CSCI method is not recommended because of adverse events (AEs) such as skin irritation. On the contrary, the CIVI method using gradual increasing ketamine minimizes AEs and is free of skin irritation. Most of hospitalized terminally ill cancer patients has proper IV access using intravascular devices (chemoport or PICC). So, CIVI method is suitable to hospitalized terminally ill cancer patients.
* This study assess the efficacy and safety of 5-days CIVI gradual dose titration of Ketamine in terminally ill cancer patients with refractory cancer pain.

ELIGIBILITY:
Inclusion Criteria:

1. Among patients with histologically or cytologically confirmed malignancy, patients with expected survival time of several months or less due to a progressive disease without additional anticancer treatment.
2. Patients with refractory cancer pain, which cases of requesting 4 or more breakthrough analgesics or increase of baseline analgesics (average pain score ≥ 4 or Personalized pain goal) in spite of 120 mg/day or more of intravenous Morphine Equivalent Daily Dose
3. Hospitalized patients with intravascular access during at least 5 days
4. Age 18 or older
5. Signed and dated informed consent of document indicating that the patient (or legally acceptable representative) has been informed about all pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

1. Patients who were treated with ketamine for pain control within 6 months
2. Patients who have been treated with radiotherapy within 4 weeks or plan to intervention for pain control during study period
3. Cancer pain cannot be excluded the Opioid induced hyperalgesia
4. Concomitant severe medical, surgical, or disease or problems which were contraindicated to application of Ketamine or have possibilities of unexpected medical problems caused be the Ketamine

   * confirmed or assumed central nervous system lesion which lead to increased intracranial pressure
   * Arrhythmia (supra-ventricular tachycardia, ventricular arrhythmia (frequent premature ventricular contraction, bigeminy, Ventricular tachycardia)
   * history of hemorrhagic stroke or seizure within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | From date of enrollment until 5 days or drop-out, assess up to 2 years
  complete pain response plus partial pain response
  * Complete pain response is defined as patient reported pain score using numerical rating scale (range 1-10) ≤ 3 or ≤ personalized pain goal (PPG) and receiving less than four rescue analgesic doses for 24 hours, without unacceptable toxicities
  * Partial pain response is defined as receiving less than four rescue analgesic doses per day without a patient reported pain score using numerical rating scale (range 1-10) ≤ 3 or ≤ personalized pain goal for 24 hr, without unacceptable toxicities

SECONDARY OUTCOMES:
Change of pain intensity | From date of enrollment until 5 days or drop-out, assess up to 2 years
  Delineate changes of pain intensity daily, from the time baseline until 5th days after application of ketamine.
  Pain intensity is defined as the mean of terdiurnal checked patient reported pain score during a day.
Rescue analgesics for breakthrough pain | From date of enrollment until 5 days or drop-out, assess up to 2 years
  Dose and number of rescue analgesics for breakthrough pain
Patient's satisfaction about Ketamine by a newly developed question in this study | at the 5th days or drop-out, assess up to 2 years
  Satisfaction about pain control and Ketamine-related distress during application of ketamine was evaluated by questions as follows: "How do you feel satisfaction about ketamine?" (at 5th days or drop-out)
Guardian's satisfaction about Ketamine by a newly developed question in this study | at the 5th days or drop-out, assess up to 2 years
  Satisfaction about pain control and Ketamine-related distress during application of ketamine was evaluated by questions as follows: "How do you feel satisfaction about ketamine?" (at 5th days or drop-out)
Rate of Ketamine-related adverse events | From date of enrollment until 5 days or drop-out, assess up to 2 years
  Rate of Ketamine-related adverse events
Rate of early discontinuation | From date of enrollment until 5 days or drop-out, assess up to 2 years
  Rate of discontinuation due to Ketamine related AEs
Overall survival | From date of enrollment until death or discharge/transfer, assess up to 2 years
  Time from application of ketamine until death or discharge/transfer

CONTACTS AND LOCATIONS:
Overall Officials: Kwonoh Park, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van den Beuken-van Everdingen MH, de Rijke JM, Kessels AG, Schouten HC, van Kleef M, Patijn J. Prevalence of pain in patients with cancer: a systematic review of the past 40 years. Ann Oncol. 2007 Sep;18(9):1437-49. doi: 10.1093/annonc/mdm056. Epub 2007 Mar 12. PMID 17355955
- [Result] Zech DFJ, Grond S, Lynch J, Hertel D, Lehmann KA. Validation of World Health Organization Guidelines for cancer pain relief: a 10-year prospective study. Pain. 1995 Oct;63(1):65-76. doi: 10.1016/0304-3959(95)00017-M. PMID 8577492
- [Result] Hanks GW, Justins DM. Cancer pain: management. Lancet. 1992 Apr 25;339(8800):1031-6. doi: 10.1016/0140-6736(92)90546-f. No abstract available. PMID 1349061
- [Result] Hardy J, Quinn S, Fazekas B, Plummer J, Eckermann S, Agar M, Spruyt O, Rowett D, Currow DC. Randomized, double-blind, placebo-controlled study to assess the efficacy and toxicity of subcutaneous ketamine in the management of cancer pain. J Clin Oncol. 2012 Oct 10;30(29):3611-7. doi: 10.1200/JCO.2012.42.1081. Epub 2012 Sep 10. PMID 22965960
- [Result] Jackson K, Ashby M, Martin P, Pisasale M, Brumley D, Hayes B. "Burst" ketamine for refractory cancer pain: an open-label audit of 39 patients. J Pain Symptom Manage. 2001 Oct;22(4):834-42. doi: 10.1016/s0885-3924(01)00340-2. PMID 11576800
- [Result] Mercadante S, Arcuri E, Tirelli W, Casuccio A. Analgesic effect of intravenous ketamine in cancer patients on morphine therapy: a randomized, controlled, double-blind, crossover, double-dose study. J Pain Symptom Manage. 2000 Oct;20(4):246-52. doi: 10.1016/s0885-3924(00)00194-9. PMID 11027905
- [Result] Bell RF, Eccleston C, Kalso EA. Ketamine as an adjuvant to opioids for cancer pain. Cochrane Database Syst Rev. 2017 Jun 28;6(6):CD003351. doi: 10.1002/14651858.CD003351.pub3. PMID 28657160
- [Derived] Park K, Kim JJ, Oh SB, Oh SY, Hong YJ, Kim SJ, Park EJ, Choi N, Shin SH, Kim S, Ko H. A Phase II Study About Efficacy and Safety of the Continuous IntraVenous Infusion of Ketamine as Adjuvant to Opioids in Terminally Ill Cancer Patients With Refractory Cancer Pain (CIVIK Trial). Am J Hosp Palliat Care. 2025 Mar;42(3):244-252. doi: 10.1177/10499091241252977. Epub 2024 May 16. PMID 38752431